CLINICAL TRIAL: NCT06012435
Title: A Randomized, Phase 3, Open-label Study to Evaluate Sigvotatug Vedotin Compared With Docetaxel in Adult Participants With Previously Treated Non-small Cell Lung Cancer (Be6A Lung-01)
Brief Title: A Study of SGN-B6A Versus Docetaxel in Previously Treated Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGNB6A-002; C5751002 (Other: Alias Study Number); 2023-503827-25-01 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-Small Lung Cancer; Seattle Genetics; lung cancer; advanced lung cancer; metastatic lung cancer; non small cell lung cancer; stage 3 lung cancer; stage 4 lung cancer; lung cancer treatment; lung cancer clinical trial; nonsquamous lung cancer; ADC; Pfizer cancer trial; vedotin; lung disease; phase 3 lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Lung Diseases | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): sigvotatug vedotin monotherapy
  Interventions: Drug: sigvotatug vedotin
- Control Arm (Active Comparator): Docetaxel monotherapy
  Interventions: Drug: docetaxel

INTERVENTIONS:
Drug: sigvotatug vedotin — Given into the vein (IV; intravenously) on Day 1 and 15 of a 28-day cycle
  Other Names: SGN-B6A; PF-08046047
  Arms: Experimental Arm
Drug: docetaxel — 75 mg/m^2 given into the vein (IV; intravenously) on Day 1 of a 21-day cycle
  Arms: Control Arm

SUMMARY:
This clinical trial is studying nonsquamous non-small cell lung cancer (NSCLC). Participants in this study must have cancer that has spread through their body or can't be removed with surgery. Participants in this study must have been treated with no more than a platinum-based chemotherapy and an anti-PD-(L)1 drug. Participants with tumors that have certain treatable genomic alterations must have had at least 1 drug for that genomic alteration, in addition to platinum-based chemotherapy.

This clinical trial uses an experimental drug called sigvotatug vedotin, which is a type of antibody drug conjugate or ADC. ADCs are designed to stick to cancer cells and kill them. This clinical trial also uses a drug called docetaxel. Docetaxel is an anticancer drug that has been approved to treat non-small cell lung cancer. It is usually given to patients who previously received another anticancer treatment. In this study, one group of participants will get sigvotatug vedotin on Days 1 and 15 during each 28-day-cycle. A second group of participants will get docetaxel on Day 1 during each 21-day cycle.

This study is being done to see if sigvotatug vedotin works better than docetaxel to treat participants with NSCLC. This study will also test what side effects happen when participants take these drugs. A side effect is anything a drug does to the body besides treating the disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of locally advanced, unresectable (Stage IIIB, IIIC), or metastatic Stage IV (M1a, M1b, or M1c) NSCLC American Joint Committee on Cancer (AJCC) Staging Manual, Version 8.0, and the Union for International Cancer Control (UICC) Staging System (Eighth edition).
* Participants must have NSCLC with nonsquamous histology

  * Tumors with squamous, or predominantly squamous histology are excluded.
  * Tumors with small cell elements are excluded.
* Participants who have NSCLC with known actionable genomic alteration (AGAs) are permitted
* Participants must have received the following prior therapies and progressed during or relapsed after receiving their most recent prior therapy:

  * Participants with no known AGAs must fulfill 1 of the following conditions:

    * Received a platinum-based combination therapy for the treatment of metastatic or recurrent disease and a PD-(L)1 monoclonal antibody (concurrently or sequentially with platinum-based chemotherapy), unless contraindicated.
    * Experienced disease progression within 6 months of the last dose of platinum-based chemotherapy in the adjuvant or neoadjuvant setting and received a PD-(L)1 monoclonal antibody at any time during the course of treatment.
  * Participants with known AGAs must fulfill the following conditions:

    * Must have received at least 1 relevant AGA targeted therapy and in the opinion of the investigator, additional AGA targeted therapy is not in the best interest of the participant.
    * Received a platinum-based combination therapy for the treatment of metastatic or recurrent disease, or experienced disease progression within 6 months of the last dose of platinum-based chemotherapy in the adjuvant or neoadjuvant setting
    * May have received up to 1 PD-(L)1 monoclonal antibody (concurrently or sequentially with platinum-based chemotherapy).
* Measurable disease based on RECIST v1.1
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, with adequate baseline hematologic, hepatic, and renal function and measurable disease according to RECIST v1.1

Exclusion Criteria:

* Life expectancy of less than (<) 3 months
* Known allergies/hypersensitivity/intolerance to or contraindication of taxanes, docetaxel, or any excipient contained in the drug formulation of sigvotatug vedotin
* History of another malignancy within 3 years before Cycle 1 Day 1, or any evidence of residual disease from a previously diagnosed malignancy. Exceptions are malignancies with a negligible risk of metastasis or death
* Participants with any of the following respiratory conditions:

  * Evidence of noninfectious interstitial lung disease (ILD) or pneumonitis that:

    * Was previous diagnosed and required systemic steroids, or
    * Is currently diagnosed and managed, or
    * Is suspected on radiologic imaging at screening
  * Known diffusing capacity of the lung for carbon monoxide (DLCO) < 50%
  * Any Grade greater than or equal to (≥) 3 pulmonary disease unrelated to underlying malignancy
* Pre-existing peripheral neuropathy Grade greater than or equal to (≥) 2
* Uncontrolled diabetes mellitus
* Prior therapy:

  * Prior treatment with antimicrotubule agents (taxanes, vinca alkaloids, or MMAEs) in the locally advanced, unresectable/refractory, or metastatic setting
  * Prior antimicrotubule agent exposure in curative settings (including adjuvant, neoadjuvant, or chemoradiotherapy) is permissible.
  * Received more than 1 prior line of cytotoxic chemotherapy in the locally advanced, unresectable/refractory, or metastatic setting
  * Prior cytotoxic chemotherapy in curative settings is permissible
  * At least 14 days must have elapsed from the last dose of radiotherapy until Cycle 1 Day 1.
  * Prior radiation therapy to the lung parenchyma that is >30 Gray (Gy) within 6 months of Cycle 1 Day 1.
  * Any systemic anticancer therapy (standard or experimental) within 21 days prior to Cycle 1 Day 1.
* Active central nervous system (CNS) lesions, including leptomeningeal metastasis, are excluded. Participants with definitively treated brain metastases are eligible in they meet the following criteria:

  * Have been clinically stable for at least 4 weeks prior to treatment initiation and baseline scans show no evidence of new or enlarged metastasis
  * On a stable dose of less than or equal to (≤) 10mg/day of prednisone or equivalent for a least 2 weeks (if requiring steroid treatment)
  * Treatment with corticosteroids greater than (>) 1 month prior to Screening visit
  * No evidence of clinical and radiographic disease progression in the CNS for ≥ 21 days after definitive radiotherapy and/or surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 703 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2026-03-12 (Estimated); Study Completion 2028-03-11 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) between the experimental arm (sigvotatug vedotin) and control arm (docetaxel) in all participants and in participants whose tumors express high levels of integrin beta-6 (IB6-high) | Approximately 5 years
  The time from date of randomization to date of death due to any cause.
Progression Free Survival (PFS) per Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) by Blinded Independent Central Review (BICR) between the experimental and control arms in all participants and in the IB6-high subgroup | Approximately 5 years
  The time from date of randomization to the first documented disease progression per RECIST v1.1 or to death due to any cause.

SECONDARY OUTCOMES:
Confirmed Objective Response Rate (ORR) per RECIST v1.1 as assessed by BICR between the experimental and control arms in all participants and in the IB6-high subgroup | Approximately 5 years
  The proportion of participants with confirmed complete response (CR) or partial response (PR) according to RECIST v1.1.
Confirmed ORR per RECIST v1.1 by investigator assessment | Approximately 5 years
  The proportion of participants with confirmed CR or PR according to RECIST v1.1.
PFS per RECIST v1.1 by investigator assessment | Approximately 5 years
  The time from date of randomization to the first documented disease progression per RECIST v1.1 or to death due to any cause.
Duration of Response (DOR) per RECIST v1.1 by BICR | Approximately 5 years
  The time from the first documented objective response (CR or PR that is subsequently confirmed) to the first documented disease progression per RECIST v1.1 or to death due to any cause.
DOR per RECIST v1.1 by investigator assessment | Approximately 5 years
  The time from the first documented objective response (CR or PR that is subsequently confirmed) to the first documented disease progression per RECIST v1.1 or to death due to any cause.
Number of participants with adverse events (AEs) | Through 30 days after the last study intervention; Approximately 5 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Mean score in the global health status/QoL combined score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | Approximately 5 years
  The EORTC QLQ-C30 was developed as a quantitative measure of health-related quality of life (HRQoL). Scores range from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/QoL represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Change from baseline in global health status/QoL combined score on the EORTC QLQ-C30 | Approximately 5 years
  The EORTC QLQ-C30 was developed as a quantitative measure of HRQoL. Scores range from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/QoL represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Mean score in physical functioning scores on the EORTC QLQ-C30 | Approximately 5 years
  The EORTC QLQ-C30 was developed as a quantitative measure of HRQoL. Scores range from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/QoL represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Change from baseline score in physical functioning scores on the EORTC QLQ-C30 | Approximately 5 years
  The EORTC QLQ-C30 was developed as a quantitative measure of HRQoL. Scores range from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/QoL represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Mean score in role functioning scores on the EORTC QLQ-C30 | Approximately 5 years
  The EORTC QLQ-C30 was developed as a quantitative measure of HRQoL. Scores range from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/QoL represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Change from baseline score in role functioning scores on the EORTC QLQ-C30 | Approximately 5 years
  The EORTC QLQ-C30 was developed as a quantitative measure of HRQoL. Scores range from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/QoL represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Mean scores in the dyspnea, cough, and chest pain scores on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer 13 (EORTC QLQ-LC13) | Approximately 5 years
  The EORTC QLQ-LC13 is a lung-cancer specific module that serves as an additional 13 item questionnaire to the general EORTC cancer questionnaire. It incorporates 1 multi-item scale to assess dyspnea, and a series of single items assessing pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis. Scores range from 0 to 100. A high score for a symptom scale/item represents a high level of symptomatology/problems.
Change from baseline in the dyspnea, cough, and chest pain scores on the EORTC QLQ-LC13 | Approximately 5 years
  The EORTC QLQ-LC13 is a lung-cancer specific module that serves as an additional 13 item questionnaire to the general EORTC cancer questionnaire. It incorporates 1 multi-item scale to assess dyspnea, and a series of single items assessing pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis. Scores range from 0 to 100. A high score for a symptom scale/item represents a high level of symptomatology/problems.
Time to Deterioration (TTD) in the global health status/QoL combined score on the EORTC QLQ-C30 | Approximately 5 years
  TTD is defined as the time from date of randomization to first onset of PRO deterioration with or without subsequent confirmation. The EORTC QLQ-C30 was developed as a quantitative measure of HRQoL. Scores range from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/QoL represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
TTD in physical functioning scores on the EORTC QLQ-C30 | Approximately 5 years
  TTD is defined as the time from date of randomization to first onset of PRO deterioration with or without subsequent confirmation. The EORTC QLQ-C30 was developed as a quantitative measure of HRQoL. Scores range from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/QoL represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
TTD in role functioning scores on the EORTC QLQ-C30 | Approximately 5 years
  TTD is defined as the time from date of randomization to first onset of PRO deterioration with or without subsequent confirmation. The EORTC QLQ-C30 was developed as a quantitative measure of HRQoL. Scores range from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/QoL represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
TTD in the dyspnea, cough, and chest pain scores on the EORTC QLQ-LC13 | Approximately 5 years
  TTD is defined as the time from date of randomization to first onset of PRO deterioration with or without subsequent confirmation. The EORTC QLQ-LC13 is a lung-cancer specific module that serves as an additional 13 item questionnaire to the general EORTC cancer questionnaire. It incorporates 1 multi-item scale to assess dyspnea, and a series of single items assessing pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis. Scores range from 0 to 100. A high score for a symptom scale/item represents a high level of symptomatology/problems.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (321):
- United States (121):
  - Alaska Oncology and Hematology, LLC, Anchorage, Alaska
  - Providence Medical Foundation, Fullerton, California
  - Providence St. Jude Medical Center Virginia K. Crosson Cancer Center and Infusion Center, Fullerton, California
  - Providence St. Jude Medical Center, Fullerton, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - Cancer Blood and Specialty Clinic, Los Alamitos, California
  - TRIO US Central Administration, Los Angeles, California
  - Drug Management Only: UCLA West Medical Pharmacy Attn: Steven L. Wong, Pharma.D., Los Angeles, California
  - Drug Management Only: UCLA West Medical Pharmacy, Attn: Steven L Wong, Pharm.D., Los Angeles, California
  - UCSF Medical Center - Mission Bay, San Francisco, California
  - Sansum Clinic, Santa Barbara, California
  - Sansum Clinic, Solvang, California
  - Rocky Mountain Cancer Centers LLP, Aurora, Colorado
  - Rocky Mountain Cancer Centers LLP, Boulder, Colorado
  - Rocky Mountain Cancer Centers LLP, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers LLP, Denver, Colorado
  - Rocky Mountain Cancer Centers LLP, Lakewood, Colorado
  - Rocky Mountain Cancer Centers LLP, Littleton, Colorado
  - Rocky Mountain Cancer Centers LLP, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers LLP, Longmont, Colorado
  - Rocky Mountain Cancer Centers LLP, Pueblo, Colorado
  - Rocky Mountain Cancer Centers LLP, Thornton, Colorado
  - Cancer Specialists of North Florida, Fleming Island, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Cancer Care Centers of Brevard, Inc., Melbourne, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - Cancer Specialists of North Florida, Neptune Beach, Florida
  - Cancer Care Centers of Brevard, Inc., Palm Bay, Florida
  - Cancer Care Centers of Brevard, Inc., Rockledge, Florida
  - Cancer Specialists of North Florida, Saint Augustine, Florida
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Maryland Oncology Hematology P.A., Annapolis, Maryland
  - Maryland Oncology Hematology P.A., Bethesda, Maryland
  - Maryland Oncology Hematology P.A., Brandywine, Maryland
  - Maryland Oncology Hematology P.A., Columbia, Maryland
  - Maryland Oncology Hematology P.A., Germantown, Maryland
  - Maryland Oncology Hematology P.A., Largo, Maryland
  - Maryland Oncology Hematology P.A., Rockville, Maryland
  - Maryland Oncology Hematology P.A., Silver Spring, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Southcoast Centers for Cancer Care, Fairhaven, Massachusetts
  - Southcoast Centers for Cancer Care, Fall River, Massachusetts
  - Allina Health Cancer Institute - Mercy Hospital, Coon Rapids, Minnesota
  - Allina Health Cancer Institute - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Allina Health Cancer Institute - United Hospital, Saint Paul, Minnesota
  - Hattiesburg Clinic Hematology/Oncology., Hattiesburg, Mississippi
  - St Luke's Cancer Institute, Kansas City, Missouri
  - Nebraska Medicine, Bellevue, Nebraska
  - Nebraska Medicine, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Summit Medical Group, Clifton, New Jersey
  - Summit Medical Group, Florham Park, New Jersey
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island, Mineola, New York
  - Laura & Isaac Perlmutter Cancer Center - NYU ACC, New York, New York
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - NYU Langone Medical Center (Tisch Hospital), New York, New York
  - University Hospitals Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - Oncology Hematology Care Clinical Trials, LLC, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center Investigational Pharmacy, Cleveland, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital Moll Cancer Pavilion, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oncology Hematology Care Clinical Trials, LLC, Fairfield, Ohio
  - Taylor Cancer Research Center, Maumee, Ohio
  - Cleveland Clinic Cancer Center/Hillcrest Hospital Cancer Center Pharmacy, Mayfield Heights, Ohio
  - University Hospitals Seidman Cancer Center at UH Mentor Health Center, Mentor, Ohio
  - UH Minoff Health Center at Chagrin Highlands, Orange, Ohio
  - Oregon Health and Science University - CHO Beaverton, Beaverton, Oregon
  - Oncology Associates of Oregon, P.C., Eugene, Oregon
  - Oregon Health and Science University - CHO Gresham, Gresham, Oregon
  - Oregon Health and Science University - CHO Northwest, Portland, Oregon
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - Oregon Health and Science University - CHO East Portland, Portland, Oregon
  - Oregon Health and Science University (CHH1), Portland, Oregon
  - Oregon Health and Science University (CHH2), Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Northwest Cancer Specialists, P.C., Tigard, Oregon
  - Oregon Health and Science University - CHO Tualatin, Tualatin, Oregon
  - Alliance Cancer Specialists, PC, Bensalem, Pennsylvania
  - Alliance Cancer Specialists, PC, Doylestown, Pennsylvania
  - Alliance Cancer Specialists, PC, Horsham, Pennsylvania
  - Alliance Cancer Specialists, PC, Langhorne, Pennsylvania
  - Alliance Cancer Specialists, PC, Media, Pennsylvania
  - Alliance Cancer Specialists, PC, Sellersville, Pennsylvania
  - Alliance Cancer Specialists, PC, Wynnewood, Pennsylvania
  - Texas Oncology - West Texas, Abilene, Texas
  - Texas Oncology - West Texas, Amarillo, Texas
  - Texas Oncology - Central South, Austin, Texas
  - University of Texas Southwestern Medical Center - Simmons Cancer Center, Dallas, Texas
  - UT Southwestern Medical Center - Redbird, Dallas, Texas
  - Univ. of TX Southwestern Medical Center - Zale Lipshy University Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center - William P. Clements, Jr., University Hospital, Dallas, Texas
  - University Of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Oncology - West Texas, El Paso, Texas
  - UT Southwestern - Simmons Cancer Center - Fort Worth, Fort Worth, Texas
  - US Oncology Investigational Product Center (IPC), Irving, Texas
  - US Oncology Investigational Products Center (IPC), Irving, Texas
  - Texas Oncology - West Texas, Midland, Texas
  - Texas Oncology - West Texas, Odessa, Texas
  - UT Southwestern - Simmons Cancer Center - Richardson/Plano, Richardson, Texas
  - Texas Oncology - Central South, Waco, Texas
  - Texas Oncology - West Texas, Wichita Falls, Texas
  - Oncology & Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Blacksburg, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, INC., Low Moor, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Roanoke, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Salem, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, INC., Wytheville, Virginia
  - Northwest Medical Specialties, PLLC, Bonney Lake, Washington
  - Northwest Medical Specialties, PLLC, Federal Way, Washington
  - Northwest Medical Specialties, PLLC, Gig Harbor, Washington
  - American Oncology Network Vista Oncology Division-West office, Olympia, Washington
  - American Oncology Network Vista Oncology Division, Olympia, Washington
  - Northwest Medical Specialties, PLLC, Puyallup, Washington
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
  - Froedtert Hospital/Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (6):
  - Instituto de Investigaciones Clinicas de Mar del Plata, Mar del Plata, Buenos Aires
  - CEMAIC - Centro Medico Privado, Córdoba, Cundinamarca
  - Sanatorio Parque, Rosario, Santa Fe Province
  - Hospital Provincial del Centenario, Rosario, Santa Fe Province
  - Sanatorio Allende Cerro, Córdoba
  - Centro Oncologico de Excelencia, San Juan
- Australia (5):
  - Border Medical Oncology Research Unit, Albury, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Peninsula Health, Frankston Hospital, Franskton, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - St John of God Hospital Murdoch, Murdoch, Western Australia
- Austria (2):
  - AKH - Medizinische Universitat Wien, Vienna
  - Riedl-Prayer-Drahanowsky-Barton Radiologiegruppenpraxis OG (RPDB)- Imagingpraterstern, Vienna
- Belgium (5):
  - Algemeen Ziekenhuis klina, Brasschaat
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Jessa Ziekenhuis VZW, Hasselt
  - CHU de Liege, Liège
- Brazil (8):
  - Oncosite - Centro de Pesquisa Clinica e Oncologia, Ijuí, Rio Grande do Sul
  - União Brasileira de Educação e Assitência (UBEA), mantenedora do Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital de Cancer de Barretos - Fundacao Pio XII, Barretos, São Paulo
  - Fundação Doutor Amaral Carvalho., Jaú, São Paulo
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia, Santo André, São Paulo
  - Centro Paulista de Oncologia S A, São Paulo, São Paulo
  - Hospital Mãe de Deus, Porto Alegre
  - Nucleo de Oncologia da Bahia - Oncoclinicas, Salvador
- Canada (11):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - William Osler Health System - Brampton Civic Hospital., Brampton, Ontario
  - William Osler Health System - Peel Memorial Hospital, Brampton, Ontario
  - William Osler Health System - Etobicoke General Hospital, Etobicoke, Ontario
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - CISSS de la Monteregie-Centre, Greenfield Park, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
- Chile (2):
  - Centro de Investigacion Clinica Bradford Hill, Recoleta, Santiago Metropolitan
  - CeCim Biocinetic, Santiago, Santiago Metropolitan
- China (29):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Fujian provincial Cancer Hospital, Fuzhou, Fujian
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Inner Mongolia Autonomous Region People's Hospital, Hothot, Inner Mongolia
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Shandong Cancer Hospital, Jinan, Shandong
  - LinYi Cancer Hospital, Linyi, Shandong
  - First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shannxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Sichuan Province Cancer Hospital, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - Beijing Chest Hospital, Capital Medical University, Beijing
  - Chongqing University Cancer Hospital, Chongqing
  - Fudan University Shanghai Cancer Center, Shanghai
- Czechia (2):
  - Vseobecna Fakultni Nemocnice v Praze, Prague, Praha 2
  - Nemocnice AGEL Ostrava Vitkovice a.s.,, Ostrava
- France (16):
  - CHU de Besancon - Hopital Jean Minjoz, Besançon
  - Centre Hospitalier de Cholet, Cholet
  - Centre Hospitalier Intercommunal Creteil - CHI Creteil, Créteil
  - CHRU de Lille, Lille
  - Hopital Nord - Batiment Mistral, Marseille
  - Centre de Cancerologie du Grand Montpellier, Montpellier
  - Service UPCC, R-1, Clinique Clementville, Montpellier
  - Hopital Cochin, APHP Centre Universite de Paris, Paris
  - Hopital Bichat-Claude Bernard - APHP, Paris
  - CHU de Bordeaux, Hopital du Haut-Leveque, Centre Francois Magendie, Pessac
  - CH de Cornouaille, Quimper
  - Centre Hospitalier Universitaire de Rennes, Hopital Pontchaillou, Rennes
  - Institut de Cancerologie Strasbourg Europe, Strasbourg
  - Hopital Sainte Musse, Toulon
  - CHU Toulouse - Hopital Larrey, Toulouse
  - IGR Gustave Roussy, Villejuif
- Germany (7):
  - Johanniter Krankenhaus Bonn, Bonn
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - Universitatsklinkik Frankfurt, Frankfurt
  - Asklepios Klinik Gauting GmbH, Gauting
  - LungenClinic Grosshansdorf, Großhansdorf
  - Krankenhaus Martha-Maria Halle Dölau gGmbH Klinik für Innere Medizin II, Halle
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
- Greece (8):
  - General Hospital of Athens Alexandra, Athens, Attikí
  - University Hospital of Larissa, Larissa, Thessaly
  - Bioiatriki Private Medical S.A., Athens
  - Henry Dunant Hospital Center, Athens
  - Metropolitan Hospital, N.Faliro
  - General University Hospital of Patras, Pátrai
  - Interbalkan Medical Center, Pilea Thessaloniki
  - St. Luke s Hospital, Thessaloniki
- Israel (5):
  - Tel Aviv Sourasky Medical Center, Tel Aviv, Other
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
- Italy (17):
  - A.O.U. - Ospedali Riuniti di Ancona, Torrette (AN), Ancona
  - Azienda Ospedaliera di Rilievo Nazionale Sant'Anna e San Sebastiano, Caserta, Campania
  - IRCCS Istituto Romagnolo per lo Studio dei Tumori Dino Amadori- IRST S.r.l, Meldola, Emilia-Romagna
  - Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Ospedale San Raffaele, Milan, Lombardy
  - Fondazione IRCCS Istituto Nazionale Dei Tumori, Milan, Lombardy
  - U.O.C. Centro di Ricerca di Fase 1, Fondazione IRCCS San Gerardo dei Tintori, Monza, MB
  - U.O.C. Oncologia Medica, Fondazione IRCCS San Gerardo dei Tintori, Monza, MB
  - Centro di Riferimento Oncologico Di Aviano, Aviano, Pordenone
  - Azienda Ospedaliera Spedali Civili di brescia, Brescia, Province OF Brescia
  - Farmacia, Roma, ROME
  - Oncologia Medica 2, Roma, ROME
  - A.O.U Policlinico G. Rodolico S. Marco, Catania, Sicily
  - G Rodolico AOU Policlinico - S. Marco, Catania
  - Clinica di Oncologia Medica Policlinico San Martino, Genova
  - UOC Oncologia Medica - Azienda Ospedaliero - Universitaria di Parma, Parma
  - Radiologia, Rome
- Japan (17):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - NHO Shikoku Cancer Center, Matsuyama, Ehime
  - Kurume University Hospital, Kurume, Fukuoka
  - Gunma Prefectural Cancer Center, Ota-Shi, Gunma
  - Kobe City Hospital Organization Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Kindai University Hospital, Sakai, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki-shi, Osaka
  - Osaka International Cancer Institute, Osaka, Other
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - Tokyo Metropolitan Cancer and Infectious diseases Center Komagome Hospital, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
- Netherlands (3):
  - Martini Ziekenhuis, Groningen
  - Maastricht UMC, Maastricht
  - Erasmus Medisch Centrum Daniel Den Hoed, Rotterdam
- Norway (4):
  - Vestre Viken Health Trust - Drammen Hospital, Drammen
  - Vestre Viken Health Trust, Drammen
  - Oslo University Hospital (OUH) - The Norwegian Radium Hospital, Oslo
  - Sykehusapoteket Oslo, Radiumhospitalet - Avdeling Produksjon, Oslo
- Poland (4):
  - Medical University of Gdansk, GdaDsk, Other
  - Instytut MSF Sp. z.o.o., Lodz
  - Institute of Genetics and Immunology GENIM LCC, Lublin
  - Med-Polonia Sp. z.o.o., Poznan
- Romania (6):
  - S.C. Medisprof S.R.L, Cluj-Napoca, Cluj
  - Ovidius Clinical Hospital, Ovidiu, Constanța County
  - Institutul Oncologic "Prof. Dr. I. Chiricuta" Cluj-Napoca, Cluj-Napoca, Koblenz
  - SC Policlinica CCBR SRL, Bucharest, Sector 3
  - Memorial Healthcare International S.R.L, Bucharest
  - Centrul de Oncologie Sf Nectarie, Craiova
- South Korea (2):
  - Ajou University Hospital., Suwon, Gyeonggi-do
  - St. Vincent's Hospital, The Catholic University of Korea., Suwon, Gyeonggido [kyonggi-do]
- Spain (16):
  - Hospital Universitario Son Espases, Palma, Balearic Islands
  - CETIR Viladomat, Barcelona, Other
  - Hospital General Universitario Alicante, Alicante, Valencia
  - Complejo Hospitalario Universitario La Coruna, A Coruña
  - Hospital General Universitario de Alicante - Farmacia, Alicante
  - lnstitut Catala D'oncologia (ICO) Badalona - Hospital Universitari Germans Trias I Pujol, Badalona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Consorcio Hospitalario Provincial de Castellon, Castellon
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Servicio de Farmacia Hospitalaria, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Quironsalud Malaga, Málaga
  - Fundación Instituto Valenciano de Oncología (FIVO), Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Clinico Universitario Lozano Blesa de Zaragoza, Zaragoza
- Switzerland (9):
  - Kantonsspital Graubuenden, Chur, Graubünden (DE)
  - Kantonsspital Graubünden/Medizinische Onkologie und Hämatologie, Chur, Graubünden (DE)
  - Universitatsspital Basel, Basel, Other
  - Kantonsspital Graubuenden, Chur, Other
  - Universitatsspital Basel, Basel
  - Inselspital, Bern
  - University Hospital Lausanne CHUV, Lausanne
  - Universitatsspital Zurich, Institut fur diagnostische und interventionelle Radiologie, Zurich
  - Universitatsspital Zurich, Zurich
- Taiwan (5):
  - National Taiwan University Hospital Yunlin Branch, Douliu, Yunlin
  - Changhua Christian Medical Foundation Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - E-Da Hospital, Kaohsiung City
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (11):
  - Diagnostic Centre, London, Others
  - The Harley Street Clinic (THSC), London, Other
  - The Royal Marsden NHS Foundation Trust (RM), Sutton, Surrey
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - St. Bartholomew's Hospital - Barts Health NHS Trust, London
  - The Royal Marsden NHS Foundation Trust (RM)., London
  - The Royal Marsden NHS Foundation Trust (RM), London
  - Sarah Cannon Research Institute UK, London
  - The Harley Street Clinic, London
  - The Christie NHS Foundation Trust, Manchester
  - Royal Marsden Hospital Sutton, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SGNB6A-002